CLINICAL TRIAL: NCT02738775
Title: A Placebo-Controlled Multi-Center Phase IIa Dose Finding Study of Ublituximab, a Third-Generation Anti-CD20 Monoclonal Antibody, in Patients With Relapsing Forms of Multiple Sclerosis.
Brief Title: Phase IIa Study of Ublituximab in Participants With Relapsing Forms of Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TG1101-RMS-201
Record Dates: First submitted 2016-04-10; First posted 2016-04-14 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ublituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1 (Experimental): Participant received intravenous (IV) infusion of ublituximab 150 milligrams (mg)/4 hour (hr) on Day 1, 450 mg/3 hr on Day 15 and 450 mg/1.5 hr on Week 24. Some participants initially received placebo IV infusion /4 hr on Day 1 and /3 hr on Day 15 before receiving ublituximab.
  Interventions: Biological: Ublituximab; Drug: Placebo
- Cohort 2 (Experimental): Participant received IV infusion of ublituximab 150 mg/4 hr on Day 1, 450 mg/1.5 hr on Day 15 and 450 mg/1 hr on Week 24. Some participants initially received placebo IV infusion /4 hr on Day 1 and /1.5 hr on Day 15 before receiving ublituximab.
  Interventions: Biological: Ublituximab; Drug: Placebo
- Cohort 3 (Experimental): Participant received IV infusion of ublituximab 150 mg/4 hr on Day 1, 450 mg/1 hr on Day 15 and 600 mg/1 hr on Week 24. Some participants initially received placebo IV infusion /4 hr on Day 1 and /1 hr on Day 15 before receiving ublituximab.
  Interventions: Biological: Ublituximab; Drug: Placebo
- Cohort 4 (Experimental): Participant received IV infusion of ublituximab 150 mg/3 hr on Day 1, 600 mg/1 hr on Day 15 and 600 mg/1 hr on Week 24. Some participants initially received placebo IV infusion /3 hr on Day 1 and /1 hr on Day 15 before receiving ublituximab.
  Interventions: Biological: Ublituximab; Drug: Placebo
- Cohort 5 (Experimental): Participant received IV infusion of ublituximab 150 mg/2 hr on Day 1, 600 mg/1 hr on Day 15 and 600 mg/1 hr on Week 24. Some participants initially received placebo IV infusion /2 hr on Day 1 and /1 hr on Day 15 before receiving ublituximab.
  Interventions: Biological: Ublituximab; Drug: Placebo
- Cohort 6 (Experimental): Participant received IV infusion of ublituximab 150 mg/1 hr on Day 1, 600 mg/1 hr on Day 15 and 600 mg/1 hr on Week 24. Some participants initially received placebo IV infusion /1 hr on Day 1 and /1 hr on Day 15 before receiving ublituximab.
  Interventions: Biological: Ublituximab; Drug: Placebo

INTERVENTIONS:
Biological: Ublituximab — Administered as an IV infusion.
  Other Names: TG-1101
Drug: Placebo

SUMMARY:
This study evaluates the use of single agent ublituximab, a novel monoclonal antibody, in participants with relapsing forms of multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing multiple sclerosis
* Active disease
* Greater than or equal to (≥) 2 relapses in prior 2 years or 1 relapse in the year prior to screening and/or ≥1 gadolinium (Gd) enhancing lesion

Exclusion Criteria:

* Treatment with anti-cluster of differentiation 20 (CD20) monoclonal antibody within the last 12 months
* Treatment with alemtuzumab within the last 12 months
* Pregnant or nursing mothers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Fox, MD, PhD, Study Chair — Central Texas Neurology
Locations (12):
- United States (12):
  - TG Therapeutics Investigational Trial Site, Phoenix, Arizona
  - TG Therapeutics Investigational Trial Site, Pasadena, California
  - TG Therapeutics Investigational Trial Site, Torrance, California
  - TG Therapeutics Investigational Trial Site, Aurora, Colorado
  - TG Therapeutics Investigational Trial Site, Fort Collins, Colorado
  - TG Therapeutics Investigational Trial Site, Lexington, Kentucky
  - TG Therapeutics Investigational Trial Site, Teaneck, New Jersey
  - TG Therapeutics Investigational Trial Site, Akron, Ohio
  - TG Therapeutics Investigational Trial Site, Columbus, Ohio
  - TG Therapeutics Investigational Trial Site, Knoxville, Tennessee
  - TG Therapeutics Investigational Trial Site, Round Rock, Texas
  - TG Therapeutics Investigational Trial Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after study completion via publication

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 49 participants were randomized in this study. One participant was treated with placebo only; 12 participants were treated with placebo prior to treatment with ublituximab.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 8 | 8 | 8 | 9 | 8 | 8
Initially Treated With Placebo | 0 | 0 | 0 | 1 | 0 | 0
Completed | 8 | 6 | 8 | 8 | 8 | 7
Not Completed | 0 | 2 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Missing | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all participants who received at least one dose of ublituximab.
Groups:
- Cohort 1: Participant received IV infusion of ublituximab 150 mg/4 hr on Day 1, 450 mg/3 hr on Day 15 and 450 mg/1.5 hr on Week 24. Some participants initially received placebo IV infusion /4 hr on Day 1 and /3 hr on Day 15 before receiving ublituximab.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.09) | 34.3 (9.13) | 44.9 (9.06) | 35.1 (9.22) | 43.5 (6.39) | 36.5 (8.33) | 39.4 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 5 | 8 | 3 | 32
  Male | 3 | 2 | 3 | 3 | 0 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 2 | 1 | 3 | 9
  Not Hispanic or Latino | 8 | 6 | 7 | 6 | 7 | 5 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 2 | 0 | 2 | 2 | 0 | 1 | 7
  Race: White | 6 | 7 | 6 | 6 | 8 | 6 | 39
  Race: Other | 0 | 1 | 0 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate of B-Cell Depletion at Week 4
Description: Responders Rate is defined as percentage of participants with greater than or equal to (≥) 95% reduction of B cells (cluster of differentiation 19 positive [CD19+] cells) within 2 weeks after the second infusion (Day 15).
Time Frame: Week 4
Population: ITT population included all participants who received at least one dose of ublituximab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
percentage of participants | 87.5 [47.35 to 99.68] | 100.0 [63.06 to 100] | 87.5 [47.35 to 99.68] | 100.0 [63.06 to 100] | 100.0 [63.06 to 100] | 100.0 [63.06 to 100]

2. Secondary Outcome: Number of New Gadolinium (Gd)-Enhancing T1 Lesions at Weeks 24 and 48
Description: The Gd-enhancing T1 lesions were evaluated using magnetic resonance imaging (MRI) technique.
Time Frame: Weeks 24 and 48
Population: ITT population included all participants who received at least one dose of ublituximab. Overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 7
lesions
  Week 24 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  Week 48 | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

3. Secondary Outcome: Number of New or Enlarging T2 Lesions at Weeks 24 and 48
Description: The new or enlarging T2 lesions were evaluated using MRI technique.
Time Frame: Weeks 24 and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- Cohort 1: Participant received IV infusion of ublituximab 150 mg/4 hr on Day 1, 450 mg /3 hr on Day 15 and 450 mg/1.5 hr on Week 24. Some participants initially received placebo IV infusion /4 hr on Day 1 and /3 hr on Day 15 before receiving ublituximab.
- Cohort 4: Participant received IV infusion of ublituximab 150 mg / 3 hr on Day 1, 600 mg / 1 hr on Day 15 and 600 mg / 1 hr on Week 24. Some participants initially received placebo IV infusion /3 hr on Day 1 and /1 hr on Day 15 before receiving ublituximab.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 7
lesions
  Week 24 | 0.38 (0.52) | 0.29 (0.49) | 0.00 (0.00) | 0.25 (0.71) | 0.00 (0.00) | 0.14 (0.38)
  Week 48 | 0.25 (0.71) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

4. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: ARR at Week 48 is calculated as the ratio of the sum of all participants confirmed relapse counts divided by the sum of all participants treatment duration (in years).
Time Frame: Week 48
Population: ITT population included all participants who received at least one dose of ublituximab.
Measure: Number; unit: relapses per participant-years
Groups:
- Cohort 4: Participant received IV infusion of ublituximab 150 mg/3 hr on Day 1, 600 mg / 1 hr on Day 15 and 600 mg/1 hr on Week 24. Some participants initially received placebo IV infusion /3 hr on Day 1 and /1 hr on Day 15 before receiving ublituximab.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
relapses per participant-years | 0.28 | 0.00 | 0.14 | 0.14 | 0.00 | 0.00

5. Secondary Outcome: Relapse Rate Reduction (RRR)
Description: RRR was calculated as the percentage reduction from baseline ARR to ARR at Week 48.
Time Frame: Baseline to Week 48
Population: ITT population included all participants who received at least one dose of ublituximab.
Measure: Number; unit: percentage reduction
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
percentage reduction | 75.55 | 100.00 | 87.80 | 89.04 | 100.00 | 100.00

6. Secondary Outcome: Percentage of Relapse Free Participants
Description: Participant was considered as free of clinical relapse if participant had no confirmed clinical relapse before treatment discontinuation/until end of Week 48. Relapses are defined as the occurrence of new or worsening neurological symptoms attributable to multiple sclerosis (MS), and immediately preceded by a stable or improving neurological state of at least 30 days.
Time Frame: Week 48
Population: ITT population included all participants who received at least one dose of ublituximab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
percentage of participants | 75.0 [34.91 to 96.81] | 100.0 [63.06 to 100] | 87.5 [47.35 to 99.68] | 87.5 [47.35 to 99.68] | 100.0 [63.06 to 100] | 100.0 [63.06 to 100]

7. Secondary Outcome: Change From Baseline in B Cells (CD19+), Memory (CD19+CD27+) and Naïve (CD19+CD27-[Negative]) B Cells
Description: Cluster of Differentiation (CD)19 is a marker of B cells, the protein has been used to diagnose cancers that arise from this type of cell - notably B cell lymphomas, acute lymphoblastic leukemia (ALL), and chronic lymphocytic leukemia (CLL). The majority of B cell malignancies express normal to high levels of CD19. Memory B cell is a type of B lymphocyte that forms part of the adaptive immune system. These cells develop within germinal centers of the secondary lymphoid organs. Their function is to memorize the characteristics of the antigen that activated their parent B cell during initial infection such that if the memory B cell later encounters the same antigen, it triggers an accelerated and robust secondary immune response. A naive B cell is a B cell that has not been exposed to an antigen. Once exposed to an antigen, the naive B cell either becomes a memory B cell or a plasma cell that secretes antibodies specific to the antigen that was originally bound.
Time Frame: Baseline, Week 1 Day 2, Week 2, Week 3 Day 15, Weeks 4, 8, 12, 16, 20, 24, Week 24 plus 2 days, Weeks 25, 28, 36, 40, 44 and 48
Population: ITT population included all participants who received at least one dose of ublituximab. 'Number analyzed' signifies participants who were evaluable for this outcome measure at the specified timepoint.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
percentage of cells
  B Cells (CD19+): Baseline | 7.40 (4.108) | 7.89 (3.899) | 7.24 (4.586) | 8.11 (2.696) | 5.71 (2.368) | 6.78 (2.097)
  B Cells (CD19+): Change from Baseline to Week 1 Day 2: number analyzed (Participants) | 8 | 7 | 7 | 8 | 8 | 8
  B Cells (CD19+): Change from Baseline to Week 1 Day 2 | -6.55 (3.920) | -8.29 (3.850) | -6.54 (4.715) | -7.95 (2.719) | -5.66 (2.347) | -6.70 (2.123)
  B Cells (CD19+): Change from Baseline to Week 2: number analyzed (Participants) | 7 | 8 | 8 | 6 | 8 | 8
  B Cells (CD19+): Change from Baseline to Week 2 | -7.52 (3.175) | -7.80 (3.878) | -7.13 (4.617) | -6.95 (1.806) | -5.68 (2.362) | -6.73 (2.090)
  B Cells (CD19+): Change from Baseline to Week 3 Day 15 | -7.27 (4.053) | -7.80 (3.830) | -7.17 (4.592) | -8.03 (2.714) | -5.69 (2.369) | -6.72 (2.080)
  B Cells (CD19+): Change from Baseline to Week 4: number analyzed (Participants) | 8 | 8 | 7 | 8 | 7 | 8
  B Cells (CD19+): Change from Baseline to Week 4 | -7.28 (4.127) | -7.79 (3.859) | -6.82 (4.889) | -8.03 (2.717) | -6.03 (2.322) | -6.71 (2.102)
  B Cells (CD19+): Change from Baseline to Week 8: number analyzed (Participants) | 8 | 8 | 8 | 7 | 8 | 8
  B Cells (CD19+): Change from Baseline to Week 8 | -7.29 (4.102) | -7.79 (3.886) | -7.15 (4.625) | -8.03 (3.032) | -5.69 (2.358) | -6.70 (2.065)
  B Cells (CD19+): Change from Baseline to Week 12: number analyzed (Participants) | 6 | 8 | 8 | 7 | 7 | 7
  B Cells (CD19+): Change from Baseline to Week 12 | -7.47 (4.592) | -7.77 (3.823) | -7.17 (4.617) | -8.45 (2.644) | -5.35 (2.317) | -7.14 (1.820)
  B Cells (CD19+): Change from Baseline to Week 16: number analyzed (Participants) | 7 | 7 | 7 | 8 | 8 | 7
  B Cells (CD19+): Change from Baseline to Week 16 | -7.01 (4.352) | -7.53 (4.110) | -7.75 (4.628) | -7.83 (2.667) | -5.68 (2.375) | -6.89 (2.178)
  B Cells (CD19+): Change from Baseline to Week 20: number analyzed (Participants) | 8 | 6 | 6 | 8 | 7 | 8
  B Cells (CD19+): Change from Baseline to Week 20 | -7.23 (4.116) | -8.07 (4.449) | -7.18 (4.637) | -7.58 (2.740) | -5.70 (2.534) | -6.65 (2.200)
  B Cells (CD19+): Change from Baseline to Week 24: number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 6
  B Cells (CD19+): Change from Baseline to Week 24 | -7.21 (4.068) | -7.53 (3.399) | -7.76 (4.478) | -7.39 (2.940) | -5.65 (2.377) | -5.62 (1.992)
  B Cells (CD19+): Change from Baseline to Week 24 Plus 2 Days: number analyzed (Participants) | 8 | 6 | 5 | 7 | 6 | 5
  B Cells (CD19+): Change from Baseline to Week 24 Plus 2 Days | -7.31 (4.108) | -6.45 (2.919) | -7.98 (4.430) | -7.88 (2.895) | -6.29 (2.403) | -7.47 (1.983)
  B Cells (CD19+): Change from Baseline to Week 25: number analyzed (Participants) | 7 | 7 | 7 | 8 | 7 | 5
  B Cells (CD19+): Change from Baseline to Week 25 | -6.45 (3.698) | -8.20 (4.007) | -7.88 (4.512) | -8.06 (2.694) | -5.57 (2.544) | -7.47 (2.008)
  B Cells (CD19+): Change from Baseline to Week 28: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 7
  B Cells (CD19+): Change from Baseline to Week 28 | -7.31 (4.106) | -6.81 (2.844) | -7.18 (4.597) | -8.00 (2.699) | -5.65 (2.360) | -6.64 (2.258)
  B Cells (CD19+): Change from Baseline to Week 36: number analyzed (Participants) | 8 | 7 | 8 | 6 | 7 | 7
  B Cells (CD19+): Change from Baseline to Week 36 | -7.32 (4.082) | -6.79 (2.820) | -7.18 (4.601) | -8.48 (2.905) | -5.69 (2.530) | -6.64 (2.255)
  B Cells (CD19+): Change from Baseline to Week 40: number analyzed (Participants) | 5 | 7 | 8 | 6 | 8 | 7
  B Cells (CD19+): Change from Baseline to Week 40 | -5.40 (3.828) | -6.74 (2.838) | -7.15 (4.567) | -7.77 (3.132) | -5.65 (2.343) | -6.56 (2.299)
  B Cells (CD19+): Change from Baseline to Week 44: number analyzed (Participants) | 8 | 7 | 8 | 7 | 8 | 7
  B Cells (CD19+): Change from Baseline to Week 44 | -7.32 (4.092) | -6.74 (2.801) | -7.05 (4.546) | -8.06 (2.860) | -5.65 (2.341) | -6.59 (2.296)
  B Cells (CD19+): Change from Baseline to Week 48: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 5
  B Cells (CD19+): Change from Baseline to Week 48 | -7.25 (4.086) | -6.71 (2.854) | -6.87 (4.542) | -7.73 (2.621) | -5.67 (2.342) | -7.39 (2.174)
  Memory (CD19+CD27+): Baseline | 0.38 (0.337) | 0.92 (0.722) | 0.90 (1.010) | 0.68 (0.457) | 0.88 (0.997) | 0.60 (0.367)
  Memory (CD19+CD27+): Change from Baseline to Week 1 Day 2: number analyzed (Participants) | 8 | 7 | 7 | 8 | 8 | 8
  Memory (CD19+CD27+): Change from Baseline to Week 1 Day 2 | -0.28 (0.279) | -0.92 (0.728) | -0.90 (1.098) | -0.59 (0.480) | -0.85 (1.001) | -0.54 (0.357)
  Memory (CD19+CD27+): Change from Baseline to Week 2: number analyzed (Participants) | 7 | 8 | 8 | 6 | 8 | 8
  Memory (CD19+CD27+): Change from Baseline to Week 2 | -0.32 (0.354) | -0.86 (0.713) | -0.83 (1.032) | -0.46 (0.411) | -0.86 (1.003) | -0.57 (0.357)
  Memory (CD19+CD27+): Change from Baseline to Week 3 Day 15 | -0.31 (0.285) | -0.86 (0.694) | -0.86 (1.007) | -0.63 (0.468) | -0.87 (1.001) | -0.57 (0.382)
  Memory (CD19+CD27+): Change from Baseline to Week 4: number analyzed (Participants) | 8 | 8 | 7 | 8 | 7 | 8
  Memory (CD19+CD27+): Change from Baseline to Week 4 | -0.31 (0.347) | -0.85 (0.690) | -0.64 (0.910) | -0.64 (0.465) | -0.91 (1.072) | -0.55 (0.396)
  Memory (CD19+CD27+): Change from Baseline to Week 8: number analyzed (Participants) | 8 | 8 | 8 | 7 | 8 | 8
  Memory (CD19+CD27+): Change from Baseline to Week 8 | -0.32 (0.331) | -0.86 (0.736) | -0.85 (1.030) | -0.64 (0.552) | -0.87 (0.994) | -0.55 (0.381)
  Memory (CD19+CD27+): Change from Baseline to Week 12: number analyzed (Participants) | 6 | 8 | 8 | 7 | 7 | 7
  Memory (CD19+CD27+): Change from Baseline to Week 12 | -0.36 (0.364) | -0.83 (0.668) | -0.87 (1.019) | -0.69 (0.494) | -0.92 (1.068) | -0.60 (0.381)
  Memory (CD19+CD27+): Change from Baseline to Week 16: number analyzed (Participants) | 7 | 7 | 7 | 8 | 8 | 7
  Memory (CD19+CD27+): Change from Baseline to Week 16 | -0.30 (0.355) | -0.92 (0.769) | -0.93 (1.068) | -0.65 (0.456) | -0.87 (1.004) | -0.56 (0.427)
  Memory (CD19+CD27+): Change from Baseline to Week 20: number analyzed (Participants) | 8 | 6 | 6 | 8 | 7 | 8
  Memory (CD19+CD27+): Change from Baseline to Week 20 | -0.27 (0.335) | -0.86 (0.849) | -1.07 (1.101) | -0.64 (0.431) | -0.88 (1.064) | -0.52 (0.421)
  Memory (CD19+CD27+): Change from Baseline to Week 24: number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 6
  Memory (CD19+CD27+): Change from Baseline to Week 24 | -0.30 (0.340) | -0.84 (0.656) | -0.96 (1.038) | -0.69 (0.442) | -0.86 (1.007) | -0.59 (0.444)
  Memory (CD19+CD27+): Change from Baseline to Week 24 Plus 2 Days: number analyzed (Participants) | 8 | 6 | 5 | 7 | 6 | 5
  Memory (CD19+CD27+): Change from Baseline to Week 24 Plus 2 Days | -0.34 (0.330) | -0.74 (0.434) | -0.76 (0.875) | -0.59 (0.469) | -0.91 (1.168) | -0.65 (0.469)
  Memory (CD19+CD27+): Change from Baseline to Week 25: number analyzed (Participants) | 7 | 7 | 7 | 8 | 7 | 6
  Memory (CD19+CD27+): Change from Baseline to Week 25 | -0.28 (0.371) | -0.97 (0.738) | -0.98 (1.057) | -0.65 (0.465) | -0.95 (1.033) | -0.61 (0.404)
  Memory (CD19+CD27+): Change from Baseline to Week 28: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 7
  Memory (CD19+CD27+): Change from Baseline to Week 28 | -0.34 (0.336) | -0.68 (0.442) | -0.87 (1.021) | -0.62 (0.508) | -0.85 (0.971) | -0.60 (0.368)
  Memory (CD19+CD27+): Change from Baseline to Week 36: number analyzed (Participants) | 8 | 7 | 8 | 6 | 7 | 7
  Memory (CD19+CD27+): Change from Baseline to Week 36 | -0.34 (0.322) | -0.68 (0.436) | -0.87 (1.020) | -0.75 (0.495) | -0.88 (1.069) | -0.59 (0.400)
  Memory (CD19+CD27+): Change from Baseline to Week 40: number analyzed (Participants) | 5 | 7 | 8 | 6 | 8 | 7
  Memory (CD19+CD27+): Change from Baseline to Week 40 | -0.20 (0.086) | -0.68 (0.441) | -0.86 (1.012) | -0.62 (0.450) | -0.85 (0.975) | -0.57 (0.424)
  Memory (CD19+CD27+): Change from Baseline to Week 44: number analyzed (Participants) | 8 | 7 | 8 | 7 | 8 | 6
  Memory (CD19+CD27+): Change from Baseline to Week 44 | -0.34 (0.341) | -0.66 (0.429) | -0.85 (0.997) | -0.69 (0.462) | -0.85 (1.008) | -0.62 (0.444)
  Memory (CD19+CD27+): Change from Baseline to Week 48: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 5
  Memory (CD19+CD27+): Change from Baseline to Week 48 | -0.32 (0.344) | -0.65 (0.463) | -0.83 (0.983) | -0.62 (0.433) | -0.86 (1.007) | -0.71 (0.414)
  Naïve (CD19+CD27-): Baseline | 6.92 (3.837) | 7.30 (3.188) | 6.26 (4.043) | 7.00 (2.135) | 4.73 (2.206) | 6.11 (2.096)
  Naïve (CD19+CD27-): Change from Baseline to Week 1 Day 2: number analyzed (Participants) | 8 | 7 | 7 | 8 | 8 | 8
  Naïve (CD19+CD27-): Change from Baseline to Week 1 Day 2 | -6.18 (3.665) | -7.29 (3.427) | -5.56 (3.954) | -6.93 (2.132) | -4.72 (2.203) | -6.09 (2.100)
  Naïve (CD19+CD27-): Change from Baseline to Week 2: number analyzed (Participants) | 7 | 8 | 8 | 6 | 8 | 8
  Naïve (CD19+CD27-): Change from Baseline to Week 2 | -7.09 (2.899) | -7.27 (3.177) | -6.23 (4.058) | -6.18 (1.723) | -4.73 (2.205) | -6.10 (2.089)
  Naïve (CD19+CD27-): Change from Baseline to Week 3 Day 15 | -6.86 (3.805) | -7.27 (3.161) | -6.23 (4.043) | -6.97 (2.137) | -4.73 (2.205) | -6.09 (2.081)
  Naïve (CD19+CD27-): Change from Baseline to Week 4: number analyzed (Participants) | 8 | 8 | 7 | 8 | 7 | 8
  Naïve (CD19+CD27-): Change from Baseline to Week 4 | -6.87 (3.836) | -7.26 (3.173) | -6.13 (4.342) | -6.96 (2.134) | -5.02 (2.211) | -6.09 (2.092)
  Naïve (CD19+CD27-): Change from Baseline to Week 8: number analyzed (Participants) | 8 | 8 | 8 | 7 | 8 | 8
  Naïve (CD19+CD27-): Change from Baseline to Week 8 | -6.88 (3.831) | -7.26 (3.173) | -6.22 (4.057) | -6.99 (2.322) | -4.73 (2.203) | -6.08 (2.093)
  Naïve (CD19+CD27-): Change from Baseline to Week 12: number analyzed (Participants) | 6 | 8 | 8 | 7 | 7 | 7
  Naïve (CD19+CD27-): Change from Baseline to Week 12 | -7.00 (4.287) | -7.26 (3.175) | -6.23 (4.061) | -7.29 (2.060) | -4.36 (2.100) | -6.47 (1.907)
  Naïve (CD19+CD27-): Change from Baseline to Week 16: number analyzed (Participants) | 7 | 7 | 7 | 8 | 8 | 7
  Naïve (CD19+CD27-): Change from Baseline to Week 16 | -6.61 (4.067) | -7.00 (3.341) | -6.74 (4.085) | -6.76 (2.098) | -4.73 (2.209) | -6.27 (2.184)
  Naïve (CD19+CD27-): Change from Baseline to Week 20: number analyzed (Participants) | 8 | 6 | 6 | 8 | 7 | 8
  Naïve (CD19+CD27-): Change from Baseline to Week 20 | -6.87 (3.828) | -7.67 (3.234) | -6.02 (3.994) | -6.52 (2.214) | -4.73 (2.377) | -6.06 (2.139)
  Naïve (CD19+CD27-): Change from Baseline to Week 24: number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 6
  Naïve (CD19+CD27-): Change from Baseline to Week 24 | -6.81 (3.788) | -7.02 (2.809) | -6.71 (4.024) | -6.26 (2.275) | -4.71 (2.207) | -4.96 (1.658)
  Naïve (CD19+CD27-): Change from Baseline to Week 24 Plus 2 Days: number analyzed (Participants) | 8 | 6 | 5 | 7 | 6 | 5
  Naïve (CD19+CD27-): Change from Baseline to Week 24 Plus 2 Days | -6.87 (3.842) | -6.18 (2.666) | -7.15 (4.231) | -6.81 (2.272) | -5.28 (2.286) | -6.74 (2.156)
  Naïve (CD19+CD27-): Change from Baseline to Week 25: number analyzed (Participants) | 7 | 7 | 7 | 8 | 7 | 5
  Naïve (CD19+CD27-): Change from Baseline to Week 25 | -6.13 (3.473) | -7.61 (3.257) | -6.81 (4.012) | -6.98 (2.132) | -4.52 (2.305) | -6.74 (2.148)
  Naïve (CD19+CD27-): Change from Baseline to Week 28: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 7
  Naïve (CD19+CD27-): Change from Baseline to Week 28 | -6.87 (3.837) | -6.53 (2.612) | -6.24 (4.047) | -6.95 (2.139) | -4.71 (2.208) | -5.97 (2.235)
  Naïve (CD19+CD27-): Change from Baseline to Week 36: number analyzed (Participants) | 8 | 7 | 8 | 6 | 7 | 7
  Naïve (CD19+CD27-): Change from Baseline to Week 36 | -6.89 (3.830) | -6.52 (2.594) | -6.23 (4.051) | -7.22 (2.249) | -4.72 (2.374) | -5.97 (2.233)
  Naïve (CD19+CD27-): Change from Baseline to Week 40: number analyzed (Participants) | 5 | 7 | 8 | 6 | 8 | 7
  Naïve (CD19+CD27-): Change from Baseline to Week 40 | -5.18 (3.740) | -6.46 (2.565) | -6.21 (4.042) | -6.63 (2.419) | -4.72 (2.204) | -5.92 (2.266)
  Naïve (CD19+CD27-): Change from Baseline to Week 44: number analyzed (Participants) | 8 | 7 | 8 | 7 | 8 | 7
  Naïve (CD19+CD27-): Change from Baseline to Week 44 | -6.89 (3.831) | -6.48 (2.573) | -6.13 (4.050) | -6.98 (2.283) | -4.72 (2.204) | -5.94 (2.248)
  Naïve (CD19+CD27-): Change from Baseline to Week 48: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 5
  Naïve (CD19+CD27-): Change from Baseline to Week 48 | -6.83 (3.809) | -6.46 (2.580) | -5.96 (4.091) | -6.69 (2.060) | -4.73 (2.205) | -6.60 (2.292)

8. Secondary Outcome: Change From Baseline in Sustained B Cell
Description: Sustained B cell reduction is defined as B-cell reductions achieved on pre-dose at Week 24 and Week 48.
Time Frame: Baseline to pre-dose at Week 24 and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
percentage of cells
  Baseline | 7.40 (4.108) | 7.89 (3.899) | 7.24 (4.586) | 8.11 (2.696) | 5.71 (2.368) | 6.78 (2.097)
  Change at Pre-dose at Week 24: number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 6
  Change at Pre-dose at Week 24 | -7.21 (4.068) | -7.53 (3.399) | -7.76 (4.478) | -7.39 (2.940) | -5.65 (2.377) | -5.62 (1.992)
  Change at Pre-dose at Week 48: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 5
  Change at Pre-dose at Week 48 | -7.25 (4.086) | -6.71 (2.854) | -6.87 (4.542) | -7.73 (2.621) | -5.67 (2.342) | -7.39 (2.174)

9. Secondary Outcome: Additional Immune Profiling-CD4+ (Cluster of Differentiation 4 Positive)
Description: A blood sample was collected and was sent to the laboratory for analysis of CD4+.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter (cells/mm^3)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
cells per cubic millimeter (cells/mm^3)
  Baseline | 28.73 (12.195) | 35.39 (4.628) | 24.34 (12.877) | 25.75 (6.874) | 22.70 (9.488) | 22.27 (10.588)
  Week 1 Day 2: number analyzed (Participants) | 8 | 7 | 7 | 8 | 8 | 8
  Week 1 Day 2 | 22.71 (15.829) | 27.52 (11.388) | 19.51 (9.129) | 16.98 (11.624) | 16.49 (13.985) | 14.15 (5.911)
  Week 2: number analyzed (Participants) | 7 | 8 | 8 | 6 | 8 | 8
  Week 2 | 34.01 (7.190) | 39.83 (8.829) | 33.31 (4.862) | 36.51 (9.289) | 28.50 (8.173) | 25.69 (8.761)
  Week 3 Day 15: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8
  Week 3 Day 15 | 23.74 (11.399) | 26.51 (10.650) | 22.60 (7.766) | 27.68 (13.656) | 19.88 (13.902) | 24.57 (11.080)
  Week 4: number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8
  Week 4 | 26.19 (11.922) | 35.31 (11.530) | 31.47 (8.658) | 30.97 (12.840) | 24.62 (8.087) | 27.59 (11.016)
  Week 8 | 29.74 (15.735) | 31.46 (8.387) | 29.64 (8.204) | 30.95 (14.625) | 27.73 (9.162) | 24.59 (4.511)
  Week 12: number analyzed (Participants) | 6 | 8 | 8 | 8 | 8 | 7
  Week 12 | 24.20 (8.152) | 32.26 (7.118) | 30.98 (11.476) | 27.71 (9.209) | 28.03 (12.045) | 24.09 (8.087)
  Week 16: number analyzed (Participants) | 7 | 7 | 7 | 8 | 8 | 7
  Week 16 | 24.03 (10.040) | 31.55 (7.557) | 19.19 (10.466) | 31.27 (12.131) | 27.37 (14.733) | 17.85 (4.155)
  Week 20: number analyzed (Participants) | 8 | 6 | 6 | 8 | 7 | 8
  Week 20 | 22.94 (9.492) | 26.87 (11.629) | 34.25 (8.928) | 33.56 (8.537) | 27.17 (7.908) | 24.51 (13.149)
  Week 24: number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 6
  Week 24 | 29.24 (8.678) | 29.36 (8.856) | 31.33 (13.406) | 29.12 (7.006) | 26.71 (9.603) | 17.41 (7.523)
  Week 24 Plus 2 Days: number analyzed (Participants) | 8 | 6 | 5 | 7 | 6 | 5
  Week 24 Plus 2 Days | 26.25 (8.120) | 27.54 (5.269) | 22.82 (17.385) | 36.47 (12.548) | 23.59 (6.912) | 21.22 (8.474)
  Week 25: number analyzed (Participants) | 7 | 6 | 7 | 8 | 7 | 5
  Week 25 | 30.70 (8.594) | 27.31 (13.091) | 35.42 (8.854) | 28.46 (9.801) | 27.96 (6.024) | 17.57 (10.438)
  Week 28: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 7
  Week 28 | 20.03 (11.870) | 31.70 (13.654) | 29.71 (13.051) | 23.57 (10.565) | 23.09 (8.855) | 21.64 (14.610)
  Week 36: number analyzed (Participants) | 8 | 7 | 8 | 7 | 7 | 7
  Week 36 | 26.79 (14.209) | 28.06 (9.436) | 37.56 (8.664) | 22.86 (8.413) | 14.73 (5.916) | 28.20 (15.386)
  Week 40: number analyzed (Participants) | 5 | 7 | 8 | 6 | 8 | 7
  Week 40 | 25.31 (10.664) | 30.91 (10.601) | 28.45 (11.497) | 28.10 (9.464) | 18.17 (11.192) | 26.68 (17.744)
  Week 44: number analyzed (Participants) | 8 | 7 | 8 | 7 | 7 | 7
  Week 44 | 24.77 (6.469) | 29.84 (9.013) | 29.83 (10.774) | 17.17 (9.920) | 26.22 (14.340) | 28.24 (12.190)
  Week 48: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 5
  Week 48 | 26.72 (6.914) | 32.92 (6.697) | 21.90 (7.779) | 22.60 (8.935) | 30.85 (13.016) | 27.03 (7.844)

10. Secondary Outcome: Additional Immune Profiling-CD8+ (Cluster of Differentiation 8 Positive)
Description: A blood sample was collected and was sent to the laboratory for analysis of CD8+.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
cells/mm^3
  Baseline | 16.80 (5.324) | 17.50 (5.222) | 9.97 (4.877) | 12.25 (2.374) | 8.72 (3.590) | 12.83 (6.576)
  Week 1 Day 2: number analyzed (Participants) | 8 | 7 | 7 | 8 | 8 | 8
  Week 1 Day 2 | 10.04 (6.698) | 12.06 (6.524) | 6.87 (2.746) | 5.93 (2.748) | 5.14 (2.779) | 7.61 (5.157)
  Week 2: number analyzed (Participants) | 7 | 8 | 8 | 6 | 8 | 8
  Week 2 | 17.03 (3.654) | 16.96 (7.869) | 13.22 (3.141) | 14.68 (2.377) | 11.14 (4.767) | 14.22 (9.157)
  Week 3 Day 15: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 8
  Week 3 Day 15 | 12.14 (6.646) | 11.88 (6.580) | 9.21 (4.780) | 12.10 (6.033) | 7.22 (4.103) | 12.50 (6.536)
  Week 4: number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8
  Week 4 | 13.89 (5.715) | 14.89 (7.815) | 11.78 (3.263) | 13.70 (5.296) | 9.89 (2.120) | 13.49 (5.214)
  Week 8 | 15.92 (8.489) | 13.91 (5.074) | 10.97 (3.012) | 12.80 (7.567) | 9.63 (3.056) | 12.62 (5.613)
  Week 12: number analyzed (Participants) | 6 | 8 | 8 | 8 | 7 | 7
  Week 12 | 15.21 (8.122) | 17.21 (6.807) | 11.83 (5.397) | 11.06 (3.773) | 8.93 (4.185) | 14.87 (9.608)
  Week 16: number analyzed (Participants) | 7 | 7 | 7 | 8 | 8 | 7
  Week 16 | 16.25 (6.951) | 13.87 (7.431) | 6.76 (3.613) | 12.51 (3.827) | 10.63 (6.203) | 10.86 (5.193)
  Week 20: number analyzed (Participants) | 8 | 6 | 6 | 8 | 7 | 8
  Week 20 | 15.04 (7.197) | 10.35 (5.998) | 10.04 (3.132) | 13.71 (3.450) | 10.29 (5.150) | 12.98 (7.476)
  Week 24: number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 6
  Week 24 | 15.83 (4.047) | 13.77 (5.509) | 11.59 (5.417) | 12.22 (5.372) | 12.05 (6.859) | 9.45 (6.093)
  Week 24 Plus 2 Days: number analyzed (Participants) | 8 | 6 | 5 | 7 | 6 | 5
  Week 24 Plus 2 Days | 14.70 (3.655) | 13.28 (6.727) | 7.05 (4.656) | 15.52 (5.839) | 8.90 (1.508) | 9.41 (3.298)
  Week 25: number analyzed (Participants) | 7 | 6 | 7 | 8 | 7 | 5
  Week 25 | 15.38 (6.717) | 12.48 (4.475) | 12.07 (4.773) | 11.60 (4.172) | 9.78 (2.395) | 8.94 (6.287)
  Week 28: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 7
  Week 28 | 11.15 (4.599) | 12.84 (5.522) | 10.63 (6.617) | 11.02 (3.030) | 9.32 (2.121) | 9.71 (3.160)
  Week 36: number analyzed (Participants) | 8 | 7 | 8 | 7 | 7 | 7
  Week 36 | 12.92 (7.721) | 11.95 (5.493) | 12.46 (2.840) | 10.11 (4.527) | 6.92 (3.158) | 11.59 (2.584)
  Week 40: number analyzed (Participants) | 5 | 7 | 8 | 6 | 8 | 7
  Week 40 | 14.63 (3.687) | 12.77 (7.654) | 9.82 (3.926) | 11.59 (4.485) | 7.93 (2.207) | 10.30 (4.027)
  Week 44: number analyzed (Participants) | 8 | 7 | 8 | 7 | 7 | 7
  Week 44 | 14.41 (6.085) | 11.46 (2.451) | 9.91 (3.937) | 8.67 (5.073) | 9.59 (3.922) | 11.87 (3.352)
  Week 48: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 5
  Week 48 | 13.28 (6.673) | 12.79 (5.232) | 7.42 (2.276) | 9.86 (5.260) | 11.68 (5.757) | 13.50 (3.412)

11. Secondary Outcome: Additional Immune Profiling-Interleukin 10 (IL10)
Description: A blood sample was collected and was sent to the laboratory for analysis of IL-10. IL-10 is an anti-inflammatory cytokine that maintains the balance of the immune response, allowing the clearance of infection while minimizing damage to the host.
Time Frame: Baseline, Weeks 2, 4, 12, 20, 24, 25, 36, 44 and 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/ml)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
picogram per milliliter (pg/ml)
  Baseline | 0.25 (0.175) | 0.37 (0.343) | 0.41 (0.459) | 0.40 (0.247) | 0.13 (0.129) | 0.09 (0.120)
  Week 2: number analyzed (Participants) | 7 | 6 | 7 | 6 | 8 | 7
  Week 2 | 0.39 (0.258) | 0.39 (0.350) | 0.27 (0.184) | 0.42 (0.070) | 0.16 (0.143) | 0.07 (0.120)
  Week 4: number analyzed (Participants) | 8 | 6 | 6 | 7 | 7 | 7
  Week 4 | 0.53 (0.294) | 0.42 (0.290) | 0.40 (0.286) | 0.34 (0.135) | 0.62 (1.059) | 0.25 (0.358)
  Week 12: number analyzed (Participants) | 5 | 7 | 8 | 8 | 7 | 7
  Week 12 | 0.57 (0.599) | 0.89 (1.223) | 0.70 (0.783) | 0.26 (0.422) | 0.04 (0.028) | 1.19 (1.147)
  Week 20: number analyzed (Participants) | 7 | 6 | 6 | 8 | 7 | 7
  Week 20 | 0.24 (0.160) | 0.65 (0.631) | 0.24 (0.141) | 0.13 (0.213) | 0.57 (0.467) | 0.64 (0.593)
  Week 24: number analyzed (Participants) | 8 | 7 | 7 | 8 | 8 | 6
  Week 24 | 0.43 (0.454) | 0.45 (0.363) | 0.49 (0.635) | 0.29 (0.325) | 2.14 (3.329) | 0.91 (0.778)
  Week 25: number analyzed (Participants) | 4 | 7 | 5 | 7 | 5 | 4
  Week 25 | 0.32 (0.163) | 0.40 (0.237) | 0.18 (0.292) | 0.24 (0.237) | 1.31 (1.168) | 1.36 (0.922)
  Week 36: number analyzed (Participants) | 7 | 7 | 8 | 7 | 7 | 6
  Week 36 | 0.21 (0.124) | 0.36 (0.543) | 0.08 (0.068) | 0.79 (0.769) | 0.95 (0.535) | 0.82 (0.303)
  Week 44: number analyzed (Participants) | 8 | 7 | 8 | 7 | 8 | 7
  Week 44 | 0.15 (0.164) | 0.35 (0.715) | 2.77 (3.101) | 1.25 (1.268) | 0.65 (0.452) | 2.11 (1.533)
  Week 48: number analyzed (Participants) | 8 | 7 | 7 | 8 | 8 | 5
  Week 48 | 0.07 (0.063) | 0.44 (0.551) | 1.87 (1.465) | 3.13 (5.552) | 0.68 (0.773) | 1.23 (0.568)

12. Secondary Outcome: Additional Immune Profiling-Natural Killer (NK) Cells
Description: A blood sample was collected and was sent to the laboratory for analysis of NK cells. Percentage of NK cells per ml of blood. NK cells are lymphocytes with the ability to kill tumor cells without deliberate immunization or activation.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of cells/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
percentage of cells/mL
  Baseline | 6.53 (2.829) | 7.22 (4.469) | 5.06 (2.618) | 7.68 (3.724) | 5.04 (2.719) | 4.67 (1.946)
  Week 1 Day 2: number analyzed (Participants) | 8 | 7 | 7 | 8 | 8 | 8
  Week 1 Day 2 | 1.98 (1.597) | 2.01 (2.465) | 2.11 (1.386) | 1.38 (0.680) | 1.10 (0.372) | 1.08 (0.980)
  Week 2: number analyzed (Participants) | 7 | 8 | 8 | 6 | 8 | 8
  Week 2 | 7.34 (6.862) | 6.03 (5.001) | 6.27 (1.230) | 7.93 (2.861) | 6.17 (3.588) | 4.09 (1.920)
  Week 3 Day 15 | 4.99 (1.647) | 6.62 (5.840) | 5.63 (2.792) | 5.93 (4.679) | 3.50 (1.717) | 4.40 (2.570)
  Week 4: number analyzed (Participants) | 8 | 8 | 7 | 8 | 7 | 8
  Week 4 | 6.45 (3.189) | 7.88 (8.131) | 7.49 (2.242) | 5.72 (2.458) | 6.12 (5.440) | 4.80 (3.352)
  Week 8: number analyzed (Participants) | 8 | 8 | 8 | 7 | 8 | 8
  Week 8 | 6.22 (4.761) | 7.53 (4.347) | 6.79 (4.172) | 4.80 (2.463) | 4.81 (2.573) | 6.21 (4.520)
  Week 12: number analyzed (Participants) | 6 | 8 | 8 | 7 | 7 | 7
  Week 12 | 5.47 (2.114) | 6.33 (3.053) | 6.71 (2.328) | 5.25 (2.494) | 3.46 (1.469) | 5.71 (2.446)
  Week 16: number analyzed (Participants) | 7 | 7 | 7 | 8 | 8 | 7
  Week 16 | 10.49 (5.747) | 5.28 (2.548) | 5.91 (3.136) | 5.34 (3.057) | 5.58 (4.578) | 7.34 (6.747)
  Week 20: number analyzed (Participants) | 8 | 6 | 6 | 8 | 7 | 8
  Week 20 | 10.17 (7.791) | 4.46 (2.638) | 6.81 (4.994) | 5.73 (2.105) | 5.79 (3.144) | 8.03 (7.391)
  Week 24: number analyzed (Participants) | 8 | 8 | 7 | 7 | 8 | 6
  Week 24 | 6.70 (4.883) | 6.51 (3.781) | 5.84 (2.890) | 4.55 (2.243) | 8.51 (5.484) | 9.81 (3.968)
  Week 24 Plus 2 Days: number analyzed (Participants) | 8 | 6 | 5 | 7 | 6 | 5
  Week 24 Plus 2 Days | 8.31 (9.513) | 4.45 (4.072) | 3.75 (2.422) | 3.38 (1.684) | 5.83 (3.711) | 4.97 (1.110)
  Week 25: number analyzed (Participants) | 7 | 7 | 7 | 8 | 7 | 5
  Week 25 | 11.45 (6.599) | 6.56 (4.849) | 5.91 (3.133) | 3.71 (2.199) | 6.51 (3.541) | 8.34 (5.602)
  Week 28: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 7
  Week 28 | 8.06 (7.674) | 5.47 (4.326) | 5.69 (3.218) | 4.73 (3.334) | 8.29 (5.664) | 6.95 (2.970)
  Week 36: number analyzed (Participants) | 8 | 7 | 8 | 6 | 7 | 7
  Week 36 | 6.63 (3.648) | 6.36 (7.256) | 5.72 (1.275) | 7.88 (5.515) | 8.22 (5.772) | 9.58 (7.535)
  Week 40: number analyzed (Participants) | 5 | 7 | 8 | 6 | 8 | 7
  Week 40 | 9.17 (4.527) | 4.67 (3.109) | 5.20 (2.904) | 6.18 (2.901) | 6.64 (3.070) | 6.90 (3.244)
  Week 44: number analyzed (Participants) | 8 | 7 | 8 | 7 | 8 | 7
  Week 44 | 7.20 (7.764) | 4.40 (3.481) | 5.00 (1.733) | 8.97 (6.008) | 6.59 (4.777) | 7.14 (3.195)
  Week 48: number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 5
  Week 48 | 3.84 (2.081) | 5.23 (4.943) | 6.72 (1.960) | 6.94 (3.601) | 7.05 (4.446) | 6.10 (1.930)

13. Secondary Outcome: Pharmacokinetic Parameter: Plasma Concentration of Ublituximab
Description: Plasma concentration is defined as the measured concentration of ublituximab.
Time Frame: Day 1 (pre-dose); Week 2; Day 15 (pre-dose); Weeks 4, 24 (pre-dose) and 25
Population: Data for this outcome measure is not reported here because as per pre-specified plan, the analysis includes pooled data from participants enrolled in multiple studies including those who were not enrolled in this study.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study medication through the end of the study (Up to 48 weeks)
Description: Safety Population included all participants who received at least one dose of ublituximab. Participants who received Placebo in any Cohort are combined for safety analysis.
Groups:
- Cohort 4: Participant received IV infusion of ublituximab 150 mg / 3 hr on Day 1, 600 mg/1 hr on Day 15 and 600 mg/1 hr on Week 24. Some participants initially received placebo IV infusion /3 hr on Day 1 and /1 hr on Day 15 before receiving ublituximab.
- Placebo: Participant received IV infusion of placebo on Day 1 and Day 15.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 2/8 | 0/8 | 0/8 | 2/8 | 0/13
Other Adverse Events (participants affected / at risk) | 8/8 | 7/8 | 8/8 | 8/8 | 8/8 | 8/8 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=8) | Cohort 3 (N=8) | Cohort 4 (N=8) | Cohort 5 (N=8) | Cohort 6 (N=8) | Placebo (N=13)
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pregnancy of partner (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=8) | Cohort 3 (N=8) | Cohort 4 (N=8) | Cohort 5 (N=8) | Cohort 6 (N=8) | Placebo (N=13)
Headache (Nervous system disorders) | 2 | 3 | 1 | 2 | 2 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 3 | 1
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 0 | 1 | 3 | 3
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Uhthoffs phenomenon (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Myelitis transverse (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vibratory sense increased (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 1 | 3 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 2 | 2 | 2 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 3 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 3 | 2 | 4 | 2 | 3 | 5
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 3 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Somnambulism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye inflammation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heart rate abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza B virus test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal odour (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT02738775/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT02738775/SAP_001.pdf